CLINICAL TRIAL: NCT00419627
Title: Proteomic Analysis of Serology and Peptides Presented on the HLA Complex of Breast, Ovarian, Colon, Rectal, Gastric and Pancreatic Adenocarcinoma.
Brief Title: Proteomic Analysis of HLA Complex in Solid Cancers: Breast, Ovary, Colon, Rectum, Stomach, and Pancreas
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Technion, Israel Institute of Technology (Other)
Other Study IDs: ProtHYMC
Record Dates: First submitted 2007-01-05; First posted 2007-01-08 (Estimated); Last update posted 2007-01-08 (Estimated); Status verified 2007-01

CONDITIONS: Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Breast Neoplasms; Ovarian Cancer
Keywords: proteomics of solid tumors
MeSH Terms: conditions — Colorectal Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to evaluate the presence of proteins in solid tumors which may lead to an immune response

DETAILED DESCRIPTION:
The main objective of the study is to evaluate which proteins are presented by the HLA complex of solid tumors. Secondary objectives include to evaluate whether an immune response specific to these proteins has actually been provoked and whether there is a similar immune response following recurrence. Real specimens will be evaluated using PCR and mass spectrometry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adenocarcinoma of breast, colon, rectum, ovary , stomach, pancreas

Exclusion Criteria:

* Withdrawal of consent
* Small specimen which does not allow to retrieve tissue without interfering with pathologic evaluation

Sex: All
Age Groups: Child, Adult, Older Adult
Enrollment: 160
Dates: Start 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Itamar Ashkenazi, M.D., Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel